CLINICAL TRIAL: NCT07154706
Title: A Phase 3 Multicenter Double-blind Randomized Study of Taletrectinib Versus Placebo in Patients With ROS1-Fusion Positive Stage IB-IIIA Non-Small Cell Lung Cancer Who Have Undergone Complete Tumor Resection
Brief Title: Phase 3 Study of Taletrectinib vs Placebo as an Adjuvant Therapy in ROS1 Positive NSCLC (TRUST-IV)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AB-106-G319
Record Dates: First submitted 2025-08-18; First posted 2025-09-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; Adjuvant; ROS1; Stage IB; Stage II; Stage IIIA; Resection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — taletrectinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Taletrectinib Active Arm (Active Comparator): Active Arm
  Interventions: Drug: Taletrectinib
- Placebo Arm (Placebo Comparator): Placebo Arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Taletrectinib — Intervention Label: Taletrectinib Intervention Name: Taletrectinib Dosage Formulation: Capsule Unit Dose Strength(s): 200 mg Dosage Level (s): 400 mg QD Route of Administration: Oral Use: Experimental IMP and NIMP/AxMP : IMP Former Name(s) or Alias(es): AB-106.
  Other Names: AB-106
  Arms: Taletrectinib Active Arm
Drug: Placebo — Intervention Label: Placebo Intervention Name: Placebo Type: Drug Dosage Formulation: Capsule Unit Dose Strength(s): 200 mg Dosage Level(s): 400 mg QD Route of Administration: Oral Use: Placebo Comparator IMP and NIMP/AxMP: IMP Former Name(s) or Alias(es): Placebo
  Arms: Placebo Arm

SUMMARY:
The purpose of this phase 3 multicenter double-blind randomized study is to assess the use of taletrectinib in the early-stage non-small cell lung cancer (NSCLC). The study compares taletrectinib (study drug) versus placebo (sugar pill) in patients with ROS1-fusion positive stage IB, II, IIIA NSCLC. The study will evaluate if taletrectinib is better than placebo at preventing the participant's disease from coming back after the participant's lung tumor was removed.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed stage IB, II, or IIIA NSCLC (AJCC 9th edition) based on pathological staging.
2. Documented ROS1 rearrangement in primary tumor by a validated local assay performed in CLIA-certified or locally equivalent diagnostic laboratories.
3. Adequate tissue is available for prospective central laboratory confirmatory testing. Confirmation of central test positivity is required prior to Randomization.

   Note: In the event that the local testing assay is the same as the central testing assay, and the local test was conducted in a CLIA-certified laboratory or local equivalent, prospective central confirmation is not needed, but tumor tissue must still be provided for other biomarker studies.
4. Age ≥18 years (or ≥20 years as required by local regulations).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Received definitive locoregional curative surgery for stage IB, II, or IIIA NSCLC. All surgical margins of resection must be negative for tumor.
7. Complete recovery from surgery (including complete wound healing) that was performed ≥4 weeks but no more than 16 weeks before Randomization if no adjuvant chemotherapy was given. Surgery must have occurred ≥4 weeks but no more than 30 weeks prior to Randomization if adjuvant chemotherapy was given. For participants who received post-resection adjuvant chemotherapy, the final dose of chemotherapy must also have occurred at least 7 days before Randomization. All chemotherapy related toxicities must have resolved to baseline or ≤Grade 1 (per CTCAE v5.0) prior to Randomization.

Exclusion Criteria:

1. Has previously received 1 or more of the following cancer treatments:

   1. Postoperative or planned radiation therapy for the current lung cancer. Note: radiotherapy in the neoadjuvant setting is allowed and must be completed at least 4 weeks prior to Randomization.
   2. Any adjuvant anticancer therapy (including investigational therapy) for treatment of NSCLC other than standard postoperative platinum-based doublet chemotherapy. Participants should have received no more than 4 cycles of the platinum doublet regimen.

      Notes: Adjuvant immune checkpoint inhibitor (ICI) treatment is allowed, but participants should have received no more than 4 cycles of the ICI, and at the time of Randomization, have at least 12 weeks of washout from the last dose of the ICI. Any prior immune-related toxicity, such as immune-related hepatitis, colitis, or pneumonitis, must be completely resolved prior to Randomization.
   3. Neoadjuvant chemotherapy with or without ICIs is allowed. Those treated with prior ICIs are eligible if ≥12 weeks have elapsed after completion of the ICI at the time of Randomization. Any prior immune-related toxicity (if an ICI was given), such as immune-related hepatitis, colitis, or pneumonitis, must be completely resolved prior to Randomization.
   4. Major surgery (including surgical resection of the primary tumor but excluding placement of vascular access port) within 4 weeks of Randomization.
   5. Segmentectomies or wedge resections, instead of complete resections, of the primary tumor. Note: These limited resections are allowed for patients with stage IB disease with T2aN0M0, with tumor size >3 to ≤4 cm, and without visceral pleura or central invasion.
2. Any investigational therapy for any condition other than NSCLC within 6 months of Randomization.
3. Co-mutations of epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) fusion.
4. History of other malignancies except adequately treated non-melanoma skin cancer, curatively treated in situ cancer, or other tumors curatively treated with no evidence of disease for >3 years after the end of treatment and which, in the opinion of the treating physician, do not have a substantial risk of recurrence of the prior malignancy.
5. Have clinically significant cardiovascular disease within 3 months prior to Randomization.
6. Have a known history of uncontrolled hypertension.
7. Experiencing ongoing cardiac dysrhythmias of ≥Grade 2 (CTCAE v5.0), uncontrolled atrial fibrillation of any CTCAE grade, a QT interval corrected by Fridericia's formula (QTcF) of >470 milliseconds, symptomatic bradycardia <45 bpm; undergoing treatment with medication(s) known to be associated with the development of Torsades de Pointes (TdP).
8. Have active and clinically significant bacterial, fungal, or viral infection, including hepatitis B virus (HBV), hepatitis C virus (HCV); or known human immunodeficiency virus (HIV)- or acquired immunodeficiency syndrome-related illness.
9. Currently have or have a history of interstitial lung disease (ILD), drug-related pneumonitis, or radiation pneumonitis that required steroid treatment.
10. Use of food or drugs that are known as strong cytochrome P450 (CYP)3A inducers or inhibitors within 14 days prior to Randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2030-08-30 (Estimated); Study Completion 2033-08-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: To compare the efficacy of taletrectinib with that of placebo, as measured by disease-free survival (DFS) by investigator assessment. | Time Frame: Up to approximately 5 years after the first patient is randomized (maximum follow-up of 70 months).
  Measure Description: Defined as the time from the date of randomization until the date of disease recurrence or death (by any cause in the absence of recurrence) by investigator's assessment.

SECONDARY OUTCOMES:
Secondary Outcome Measure: DFS rates by investigator assessment at 2, 3, 4, and 5 years. | Time Frame: Up to approximately 5 years after the first patient is randomized (maximum follow-up of 70 months). DFS rate 2 years (%), 3 years (%), 4 years (%), and 5 years (%) are presented.
  Measure Description: The percentage of participants disease free and alive as determined by investigator assessment at 2, 3, 4, and 5 years after date of randomization.
Secondary Outcome Measure: Overall Survival (OS). | Time Frame: Up to approximately 7 years after the first patient is randomized (maximum follow-up of 86 months).
  Measure Description: Defined as the time from the date of randomization until date of death due to any cause.
Secondary Outcome Measure: DFS by blinded independent central review (BICR). | Time Frame: Up to approximately 5 years after the first patient is randomized (maximum follow-up of 70 months).
  Measure Description: Defined as the time from the date of randomization until the date of disease recurrence of death (by any cause in the absence of recurrence) by blinded independent central review.
Secondary Outcome Measure: OS rates at 2, 3, 4, and 5 years. | Time Frame: Up to approximately 7 years after the first patient is randomized (maximum follow-up of 86 months). DFS rate 2 years (%), 3 years (%), 4 years (%), and 5 years (%) are presented.
  Measure Description: The percent of participants that are alive at 2, 3, 4, and 5 years after date of randomization.
Secondary Outcome Measure: Central nervous system (CNS) DFS by Investigator assessment and by BICR. | Time Frame: Up to approximately 5 years after the first patient is randomized (maximum follow-up of 70 months).
  Measure Description: Defined as the time from the date of randomization until the date of disease recurrence within the CNS or death (by any cause in the absence of recurrence) by investigator's assessment and blinded independent central review.
Secondary Outcome Measure: Plasma concentrations of taletrectinib. | Time Frame: Collected between 1-3 hours post-dose on Cycle1 Day 1, and pre-dose and 1-3 hours post-dose at Cycle 2 Day 1, and pre-dose at Cycle 4 Day 1, and Cycle 7 Day 1. The length of each cycle is 28 days.
  Measure Description: The pharmacokinetics exposure parameters derived from plasma concentrations of taletrectinib.
Secondary Outcome Measure: Incidence of adverse events (AEs). | Time Frame: Up to approximately 5 years after the first patient is randomized (maximum follow-up of 70 months).
  Measure Description: Defined as the number of patients reporting adverse events within one study arm compared to the overall number of patients within the same study arm.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - UCLA, Los Angeles, California
  - Georgetown University Medical Cener (GUMC), Washington D.C., District of Columbia
  - Saint Alphonsus Health System, Boise, Idaho
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute (SCRI) - Texas Oncology-Central South, Austin, Texas
  - MD Anderson, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Princess Margaret Cancer Centre-University Health Network, Toronto, Ontario, Canada